CLINICAL TRIAL: NCT01004562
Title: The Breast Cancer Specialized Program of Research Excellence (SPORE): Core A-Administrative/Biostatistics Core
Brief Title: Collecting Information From Patients Enrolled in the Breast Specialized Program of Research Excellence
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000378061; UAB-X010112005
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: informational intervention

SUMMARY:
RATIONALE: Collecting and storing information from patients with cancer to study in the future may help doctors learn more about cancer.

PURPOSE: This study is collecting information from patients enrolled in the Breast Specialized Program of Research Excellence.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide a database for administrative and biostatistical support for the Breast Specialized Program of Research Excellence.

OUTLINE: Data is collected from patients for future research studies.

PROJECTED ACCRUAL: A total of 535 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer patients of any age
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2007-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Administrative and biostatistical support for the Breast Specialized Program of Research Excellence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yufeng Li, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Comprehensive Cancer Center, Birmingham, Alabama, United States